CLINICAL TRIAL: NCT05730803
Title: Study on the Displacement of Iodine Balance Value During Pregnancy and the Mechanism of Breast Iodine Homeostasis During Lactation Under Different Iodine Exposure
Brief Title: Displacement of Iodine Balance Value During Pregnancy and the Mechanism of Breast Iodine Homeostasis During Lactation
Status: Not yet recruiting | Type: Observational
Sponsor: Tianjin Medical University (Other)
Responsible Party: Principal Investigator, Wanqi Zhang, professor, Tianjin Medical University
Other Study IDs: NSFC-8223000919
Record Dates: First submitted 2023-02-02; First posted 2023-02-16 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Nutritional Requirements
Keywords: nutrition of special population; nutrient; trace element iodine; zero balance displacement; large variation of breastmilk
MeSH Terms: interventions — Diet Therapy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — blood, urine, breast milk, faeces
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: dietary intervention — During the iodine balance period of pregnant women, seaweed was added to lunch on the 4-6 days of the experiment, and the iodine content was about 200 μg.

SUMMARY:
In order to solve the bottleneck problems of"zero balance displacement"and"large variation of breastmilk"in the study of iodine EAR of pregnant women, lactating women and infants, firstly, this study intends to clarify the rate of metabolism and distribution of iodine during pregnancy by 125I tracer, SPECT/CT in vivo small animal imaging and γ counting study. Then, the iodine balance study in rats was conducted to verify the degree of "zero balance value displacement"caused by the difference of iodine absorption and store in different organs and tissues under different iodine exposure levels, so as to determine the iodine selection conditions of subjects in the population experiment. To determine the EAR of pregnant women by optimizing the population iodine balance experiment. Secondly, we proposed to study the regulatory mechanism of NIS and Pendrin in the mammary gland of lactating rats under different iodine nutrition levels to clarify the range of breastmilk iodine compensation. Mammary cell experiments intend to clarify the mutual regulations of iodine nutrition, oestrogen, and NIS and Pendrin. Based on the results of animal and cellular experiments, and the effect of genetic, oestrogen and iodine status were considered, a cross-sectional study of lactating women was conducted to determine the normal reference range of breastmilk iodine after screening out the people with abnormal indicators. This study will solve the bottleneck problems and difficulties in the iodine RNI research for pregnant women, lactating women and infants, found the iodine nutritional compensatory mechanism under special physiology, and provide the scientific basis for obtaining the accurate EAR basic data and the revision of iodine DRIs.

DETAILED DESCRIPTION:
In this study, the absorption, distribution, storage and excretion of 125I in rats were observed by small animal imaging technology in vivo, so as to clarify the characteristics of iodine metabolism under different iodine exposure, and provide a basis for optimizing the experimental cycle of iodine balance experiment. The iodine balance experiment of rats during pregnancy was carried out, the iodine storage in different organs was detected to explain the phenomenon of "zero point balance value shift", and the population with iodine nutrition background was determined as the experimental objects in the iodine balance experiment. The optimized iodine balance experiment was further verified in the population, and the iodine EAR of pregnant women was explored to provide reference data for formulating the recommended iodine intake of pregnant women in China in the future. The expression difference of NIS and Pendrin in lactating rats with different iodine nutritional status was used to determine the range of milk iodine compensation. To determine the synergistic and independent effects of iodine level and estrogen on the expression of NIS and Pendrin in lactating mammary gland cells cultured in primary culture. Through a cross-section study of lactating women, the correlation between milk iodine level and NIS, Pendrin gene mutation, iodine exposure level and estrogen was discussed, the phenomenon of "huge milk iodine variation" was explained, the normal reference range of milk iodine was defined, and the basis was laid for further determination of iodine AI and EAR of lactating mothers in 0-6 months. To clarify the steady-state mechanism of iodine metabolism in pregnancy-milk during special physiological periods with different iodine exposure levels, research ideas and related research results can also provide references for the determination of other nutrient requirements.

ELIGIBILITY:
Inclusion Criteria:

Pregnant women:

* Aged 18-40, who have lived in the area for ≥5 year;
* Single pregnancy;
* Those who have no special dietary habits;

Lactating woman:

* Breastfeeding a child;
* Normal thyroid function during pregnancy;
* Term delivery (38-42 weeks of gestation);

Exclusion Criteria:

Pregnant women:

* Smoking or drinking;
* Iodized drugs or contrast agents have been used in the past year;
* A history of thyroid disease, autoimmune disease, endocrine disease, heart disease, chronic disease or family hereditary disease, etc

Lactating woman:

* A history of thyroid disease, autoimmune disease, endocrine disease, heart disease, chronic disease or family hereditary disease, etc;
* Iodized drugs or contrast agents have been used;

Ages: 1 Day to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Women in the third trimester (18-40 years old), lactating women (38-42 weeks of gestation), all from Tianjin, Xinjiang and Gansu.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2023-02-17 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
urine iodine concentration | pregnancy 1-40 weeks
  μg/L
Free thyroxine | pregnancy 1-40 weeks
  pmol/L
Free triiodothyronine | pregnancy 1-40 weeks
  pmol/L
Thyroglobulin(TG) | pregnancy 1-40 weeks
  ug/L
Thyroid-stimulating hormone | pregnancy 1-40 weeks
  mIU/L
Salt iodine concentration | pregnancy 1-40 weeks
  μg/day
Urinary iodine excretion | pregnancy 1-40 weeks
  μg/day
Fecal iodine excretion | pregnancy 1-40 weeks
  μg/day
Dietary iodine intake | pregnancy 1-40 weeks
  μg/day
Water iodine intake | pregnancy 1-40 weeks
  ug/day
Thyroid peroxidase antibody | pregnancy 1-40 weeks
  IU/mL
Thyroglobulin antibody | pregnancy 1-40 weeks
  IU/mL
Milk iodine excretion | Postpartum 0-6 months
  μg/day
Milk Iodine concentration | Postpartum 0-6 months
  μg/L
Thyroid volume | Postpartum 0-6 months
  cm³
Na+/I- symporter | Postpartum 0-6 months
  mRNA
Pendrin | Postpartum 0-6 months
  mRNA
estrogen | Postpartum 0-6 months
  pmol/L
progesterone | Postpartum 0-6 months
  pmol/L
oxytocin | Postpartum 0-6 months
  ng/L
prolactin | Postpartum 0-6 months
  pg/MI

SECONDARY OUTCOMES:
Milk output | Postpartum 0-6 months
  μg/day

CONTACTS AND LOCATIONS:
Overall Officials: Ling Zhang, Principal Investigator — Xinjiang Uygur Autonomous Region Center for Disease Control and Prevention; Yanling Wang, Principal Investigator — Gansu Provincial Center for Disease Control and Prevention; Xiaomei Yao, Principal Investigator — Tianjin Medical University; Laixiang Lin, Principal Investigator — Tianjin Medical University; Zuoliang Dong, Principal Investigator — Tianjin Medical University; Yiming Shen, Principal Investigator — Tianjin Medical University; Chenchen Wang, Principal Investigator — Xinjiang Uygur Autonomous Region Center for Disease Control and Prevention; Wenxing Guo, Principal Investigator — Tianjin Medical University; Ziyun Pan, Principal Investigator — Tianjin Medical University
Locations (2):
- China (2):
  - Gansu Provincial Center for Disease Control and Prevention, Lanzhou
  - Xinjiang Uygur Autonomous Region Center for Disease Control and Prevention, Ürümqi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stinca S, Andersson M, Herter-Aeberli I, Chabaa L, Cherkaoui M, El Ansari N, Aboussad A, Weibel S, Zimmermann MB. Moderate-to-Severe Iodine Deficiency in the "First 1000 Days" Causes More Thyroid Hypofunction in Infants Than in Pregnant or Lactating Women. J Nutr. 2017 Apr;147(4):589-595. doi: 10.3945/jn.116.244665. Epub 2017 Feb 15. PMID 28202636
- [Background] Gao M, Chen W, Sun H, Fan L, Wang W, Du C, Chen Y, Lin L, Pearce EN, Shen J, Cheng Y, Wang C, Zhang W. Excessive iodine intake is associated with formation of thyroid nodules in pregnant Chinese women. Nutr Res. 2019 Jun;66:61-67. doi: 10.1016/j.nutres.2019.02.009. Epub 2019 Mar 6. PMID 30979661
- [Background] Pearce EN, Lazarus JH, Moreno-Reyes R, Zimmermann MB. Consequences of iodine deficiency and excess in pregnant women: an overview of current knowns and unknowns. Am J Clin Nutr. 2016 Sep;104 Suppl 3(Suppl 3):918S-23S. doi: 10.3945/ajcn.115.110429. Epub 2016 Aug 17. PMID 27534632
- [Background] Sang Z, Wang PP, Yao Z, Shen J, Halfyard B, Tan L, Zhao N, Wu Y, Gao S, Tan J, Liu J, Chen Z, Zhang W. Exploration of the safe upper level of iodine intake in euthyroid Chinese adults: a randomized double-blind trial. Am J Clin Nutr. 2012 Feb;95(2):367-73. doi: 10.3945/ajcn.111.028001. Epub 2011 Dec 28. PMID 22205314
- [Background] Chen W, Li X, Wu Y, Bian J, Shen J, Jiang W, Tan L, Wang X, Wang W, Pearce EN, Zimmermann MB, Carriquiry AL, Zhang W. Associations between iodine intake, thyroid volume, and goiter rate in school-aged Chinese children from areas with high iodine drinking water concentrations. Am J Clin Nutr. 2017 Jan;105(1):228-233. doi: 10.3945/ajcn.116.139725. Epub 2016 Dec 7. PMID 27927635
- [Background] Chen W, Zhang Y, Hao Y, Wang W, Tan L, Bian J, Pearce EN, Zimmermann MB, Shen J, Zhang W. Adverse effects on thyroid of Chinese children exposed to long-term iodine excess: optimal and safe Tolerable Upper Intake Levels of iodine for 7- to 14-y-old children. Am J Clin Nutr. 2018 May 1;107(5):780-788. doi: 10.1093/ajcn/nqy011. PMID 29722836
- [Background] Sang Z, Wei W, Zhao N, Zhang G, Chen W, Liu H, Shen J, Liu J, Yan Y, Zhang W. Thyroid dysfunction during late gestation is associated with excessive iodine intake in pregnant women. J Clin Endocrinol Metab. 2012 Aug;97(8):E1363-9. doi: 10.1210/jc.2011-3438. Epub 2012 Jun 5. PMID 22669304
- [Background] Shi X, Han C, Li C, Mao J, Wang W, Xie X, Li C, Xu B, Meng T, Du J, Zhang S, Gao Z, Zhang X, Fan C, Shan Z, Teng W. Optimal and safe upper limits of iodine intake for early pregnancy in iodine-sufficient regions: a cross-sectional study of 7190 pregnant women in China. J Clin Endocrinol Metab. 2015 Apr;100(4):1630-8. doi: 10.1210/jc.2014-3704. Epub 2015 Jan 28. PMID 25629356
- [Background] Yang L, Li M, Liu X, Wu M, Zhang J, Zhao L, Ding G, Yang X. Evaluation of Iodine Nutritional Status Among Pregnant Women in China. Thyroid. 2020 Mar;30(3):443-450. doi: 10.1089/thy.2019.0001. PMID 31964276
- [Background] Tan L, Tian X, Wang W, Guo X, Sang Z, Li X, Zhang P, Sun Y, Tang C, Xu Z, Shen J, Zhang W. Exploration of the appropriate recommended nutrient intake of iodine in healthy Chinese women: an iodine balance experiment. Br J Nutr. 2019 Mar 14;121(5):519-528. doi: 10.1017/S0007114518003653. Epub 2018 Dec 11. PMID 30526700
- [Background] Andersson M, Braegger CP. The Role of Iodine for Thyroid Function in Lactating Women and Infants. Endocr Rev. 2021 Nov 17:bnab029. doi: 10.1210/endrev/bnab029. Online ahead of print. Erratum In: Endocr Rev. 2022 May 12;43(3):610. PMID 34791141
- [Background] Stravik M, Gustin K, Barman M, Skroder H, Sandin A, Wold AE, Sandberg AS, Kippler M, Vahter M. Infant Iodine and Selenium Status in Relation to Maternal Status and Diet During Pregnancy and Lactation. Front Nutr. 2021 Dec 17;8:733602. doi: 10.3389/fnut.2021.733602. eCollection 2021. PMID 34988107
- [Background] Zimmermann MB. The adverse effects of mild-to-moderate iodine deficiency during pregnancy and childhood: a review. Thyroid. 2007 Sep;17(9):829-35. doi: 10.1089/thy.2007.0108. PMID 17956157
- [Background] Naess S, Markhus MW, Strand TA, Kjellevold M, Dahl L, Stokland AM, Nedrebo BG, Aakre I. Iodine Nutrition and Iodine Supplement Initiation in Association with Thyroid Function in Mildly-to-Moderately Iodine-Deficient Pregnant and Postpartum Women. J Nutr. 2021 Oct 1;151(10):3187-3196. doi: 10.1093/jn/nxab224. PMID 34255063
- [Background] Zhang H, Wu M, Yang L, Wu J, Hu Y, Han J, Gu Y, Li X, Wang H, Ma L, Yang X. Evaluation of median urinary iodine concentration cut-off for defining iodine deficiency in pregnant women after a long term USI in China. Nutr Metab (Lond). 2019 Sep 9;16:62. doi: 10.1186/s12986-019-0381-4. eCollection 2019. PMID 31516542
- [Background] Dold S, Zimmermann MB, Baumgartner J, Davaz T, Galetti V, Braegger C, Andersson M. A dose-response crossover iodine balance study to determine iodine requirements in early infancy. Am J Clin Nutr. 2016 Sep;104(3):620-8. doi: 10.3945/ajcn.116.134049. Epub 2016 Jul 27. PMID 27465383
- [Background] Semba RD, Delange F. Iodine in human milk: perspectives for infant health. Nutr Rev. 2001 Aug;59(8 Pt 1):269-78. doi: 10.1111/j.1753-4887.2001.tb05512.x. PMID 11518182
- [Background] Nazeri P, Mirmiran P, Shiva N, Mehrabi Y, Mojarrad M, Azizi F. Iodine nutrition status in lactating mothers residing in countries with mandatory and voluntary iodine fortification programs: an updated systematic review. Thyroid. 2015 Jun;25(6):611-20. doi: 10.1089/thy.2014.0491. Epub 2015 May 14. PMID 25811835
- [Background] Chen Y, Gao M, Bai Y, Hao Y, Chen W, Cui T, Guo W, Pan Z, Lin L, Wang C, Shen J, Zhang W. Variation of iodine concentration in breast milk and urine in exclusively breastfeeding women and their infants during the first 24 wk after childbirth. Nutrition. 2020 Mar;71:110599. doi: 10.1016/j.nut.2019.110599. Epub 2019 Sep 23. PMID 31901706
- [Background] Azizi F, Smyth P. Breastfeeding and maternal and infant iodine nutrition. Clin Endocrinol (Oxf). 2009 May;70(5):803-9. doi: 10.1111/j.1365-2265.2008.03442.x. Epub 2008 Oct 6. PMID 19178515
- [Background] Dold S, Zimmermann MB, Aboussad A, Cherkaoui M, Jia Q, Jukic T, Kusic Z, Quirino A, Sang Z, San Luis TO, Vandea E, Andersson M. Breast Milk Iodine Concentration Is a More Accurate Biomarker of Iodine Status Than Urinary Iodine Concentration in Exclusively Breastfeeding Women. J Nutr. 2017 Apr;147(4):528-537. doi: 10.3945/jn.116.242560. Epub 2017 Feb 22. PMID 28228508
- [Background] Yang L, Wang J, Yang J, Zhang H, Liu X, Mao D, Lu J, Gu Y, Li X, Wang H, Xu J, Tan H, Zhang H, Yu W, Tao X, Fan Y, Cai Q, Liu X, Yang X. An iodine balance study to explore the recommended nutrient intake of iodine in Chinese young adults. Br J Nutr. 2020 Dec 14;124(11):1156-1165. doi: 10.1017/S0007114520002196. Epub 2020 Jun 22. PMID 32624007
- [Background] Dworkin HJ, Jacquez JA, Beierwaltes WH. Relationship of iodine ingestion to iodine excretion in pregnancy. J Clin Endocrinol Metab. 1966 Dec;26(12):1329-42. doi: 10.1210/jcem-26-12-1329. No abstract available. PMID 5959526
- [Background] Teng D, Yang W, Shi X, Li Y, Ba J, Chen B, Du J, He L, Lai X, Li Y, Chi H, Liao E, Liu C, Liu L, Qin G, Qin Y, Quan H, Shi B, Sun H, Tang X, Tong N, Wang G, Zhang JA, Wang Y, Xue Y, Yan L, Yang J, Yang L, Yao Y, Ye Z, Zhang Q, Zhang L, Zhu J, Zhu M, Shan Z, Teng W. An Inverse Relationship Between Iodine Intake and Thyroid Antibodies: A National Cross-Sectional Survey in Mainland China. Thyroid. 2020 Nov;30(11):1656-1665. doi: 10.1089/thy.2020.0037. Epub 2020 Jul 23. PMID 32586221
- [Background] Lee YA, Cho SW, Sung HK, Kim K, Song YS, Moon SJ, Oh JW, Ju DL, Choi S, Song SH, Cheon GJ, Park YJ, Shin CH, Park SK, Jun JK, Chung JK. Effects of Maternal Iodine Status during Pregnancy and Lactation on Maternal Thyroid Function and Offspring Growth and Development: A Prospective Study Protocol for the Ideal Breast Milk Cohort. Endocrinol Metab (Seoul). 2018 Sep;33(3):395-402. doi: 10.3803/EnM.2018.33.3.395. PMID 30229579
- [Background] Rillema JA, Hill MA. Prolactin regulation of the pendrin-iodide transporter in the mammary gland. Am J Physiol Endocrinol Metab. 2003 Jan;284(1):E25-8. doi: 10.1152/ajpendo.00383.2002. Epub 2002 Sep 11. PMID 12388138
- [Background] Dror DK, Allen LH. Iodine in Human Milk: A Systematic Review. Adv Nutr. 2018 May 1;9(suppl_1):347S-357S. doi: 10.1093/advances/nmy020. PMID 29846524
- [Background] Kennett JE, Poletini MO, Fitch CA, Freeman ME. Antagonism of oxytocin prevents suckling- and estradiol-induced, but not progesterone-induced, secretion of prolactin. Endocrinology. 2009 May;150(5):2292-9. doi: 10.1210/en.2008-1611. Epub 2008 Dec 23. PMID 19106214
- [Background] Mizokami T, Fukata S, Hishinuma A, Kogai T, Hamada K, Maruta T, Higashi K, Tajiri J. Iodide Transport Defect and Breast Milk Iodine. Eur Thyroid J. 2016 Jul;5(2):145-8. doi: 10.1159/000446496. Epub 2016 May 27. PMID 27493890
- [Background] Al-Rasheed MM, Alzahrani AS, Macadam A, Overall A, Gard P, Dzimiri N. The potential role of the sodium iodide symporter gene polymorphism in the development of differentiated thyroid cancer. Gene. 2015 Nov 10;572(2):163-8. doi: 10.1016/j.gene.2015.07.009. Epub 2015 Jul 6. PMID 26160439